CLINICAL TRIAL: NCT00853632
Title: Carpentier-Edwards® Perimount Magna® Mitral Pericardial Bioprostheses Models 7000/7000 TFX and Carpentier-Edwards® Perimount Magna® Mitral Ease™ Pericardial Bioprostheses Models 7200TFX and 7300/7300TFX
Brief Title: Magna® Mitral Pericardial Bioprostheses Post-Approval Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-05
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease; Mitral Valve Regurgitation; Mitral Valve Incompetence; Heart Failure
Keywords: Mitral valve; pericardial bioprostheses; PERIMOUNT; bovine pericardial leaflets; mitral valve replacement; mitral valve regurgitation; Heart valve disease
MeSH Terms: conditions — Coronary Artery Disease; Mitral Valve Insufficiency; Heart Failure; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Device - CEP Mitral Valve (Other)
  Interventions: Device: CEP MAGNA MITRAL PERICARDIAL BIOPROSTHESES

INTERVENTIONS:
Device: CEP MAGNA MITRAL PERICARDIAL BIOPROSTHESES — Mitral valve replacement
  Other Names: Magna Mitral 7000/7000TFX, Magna Mitral Ease 7200TFX, 7300/7300TFX

SUMMARY:
The purpose of the study is to demonstrate the long term safety and effectiveness of the Carpentier-Edwards® PERIMOUNT Magna Mitral Valves in patients undergoing mitral valve replacement with or without concomitant procedures requiring cardiopulmonary bypass.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center study to be conducted in the US and outside the US (OUS). Approximately 250 subjects are planned to be enrolled to obtain long term data from 101 subjects at 8 years post implant of the Magna mitral valve. Of these 250, approximately 38 (15%) are anticipated to be simultaneous aortic and mitral replacements. Subject enrollment will not start in the US before obtaining FDA approval of this post market study.

Assessments will be obtained for the preoperative and operative visits, and postoperatively at discharge, six months, 1-year and annually thereafter for a minimum of 8 years. Subject's demographics (date of birth, sex), physical assessment (heart rate, height, weight, systolic and diastolic blood pressures), New York Heart Association (NYHA) functional class, cardiac rhythm, cardiovascular medical history/risk factors, non-cardiovascular conditions, previous cardiovascular procedures/interventions, antithromboembolic and lipid lowering medications and coagulation profile. Blood data will be collected from each subject preoperatively, at 6 months and annually post implant through 8 year follow-ups. Echocardiographic evaluation required for each subject preoperatively, at discharge, 6 months (between 3-6 months), 1, 2, 4, 6, and 8 year follow-ups. A QOL survey (EQ-5D) will be completed by the subject pre-operatively and at the 6-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* The patient requires, as indicated in the preoperative evaluation, a replacement mitral valve.
* The patient has signed and dated the subject informed consent form prior to surgery.
* The patient is expected to survive the surgery and be discharged.
* The patient is geographically stable and agrees to attend follow-up assessments.
* The patient is 18 years or older.

Exclusion Criteria:

* The patient has any known non-cardiac life-threatening disease, which will limit the patient's life expectancy below 1 year.
* The patient presents with active endocarditis within the last 3 months.
* The patient is pregnant or lactating.
* The patient is an intravenous drug abuser.
* The patient is currently a prison inmate.
* The patient is currently participating in a study of an investigational drug or device.
* The patient requires replacement of a native or prosthetic tricuspid or pulmonic valve.
* The patient requires replacement of a native or prosthetic aortic valve with a prosthesis other than a commercially available Carpentier-Edwards PERIMOUNT Valve (i.e. models 2700, 2700TFX, 2800, 2800TFX, 2900, 3000, 3000TFX, 3300TFX)*.
* The patient was previously enrolled in the study.
* The patient has had prior aortic, tricuspid and/or pulmonary valve surgery, which included implantation of a bioprosthetic valve or mechanical valve that will remain in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2007-08; Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (10):
  - Dignity Health Research Institute, Sacramento, California
  - AdventHealth Orlando, Orlando, Florida
  - Northwestern University Hospital, Chicago, Illinois
  - University of Iowa Hospital & Clinics, Iowa City, Iowa
  - Iowa Heart Medical Center, West Des Moines, Iowa
  - University of Michigan Medical School, Ann Arbor, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Missouri Baptist Medical Center, St Louis, Missouri
  - North Shore University Hospital, NY, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
- Krankenhaus Hietzing, Vienna, Austria
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Germany (2):
  - University Clinica Eppendorf, Hamburg
  - Klinikum der Friedrich Schiller University, Jena

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Device - CEP Mitral Valve: Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve
Period: Overall Study
Arm/Group | Device - CEP Mitral Valve
Started | 329
Completed | 127
Not Completed | 202
Not completed — Death | 88
Not completed — Withdrawal by Subject | 45
Not completed — Lost to Follow-up | 30
Not completed — Reoperation/Explant | 17
Not completed — Exit with other reason | 22

BASELINE CHARACTERISTICS:
Population: Subjects implanted with a Carpentier-Edwards PERIMOUNT Magna Mitral heart valve.
Groups:
- Device - CEP Mitral Valve: Subjects who received a Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 329
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201
  Male | 128
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 55
  Europe | 105
  United States | 169

OUTCOME MEASURES:

1. Primary Outcome: Subject's Rate of Objective Performance Criteria Per ISO 5840-2005 - Total Number of Late Adverse Events (by Category) Divided by Late Patient Years (Expressed as a Percentage) for the Magna Mitral Valve Implanted Cohort
Description: A linearized rate percentage is calculated by the following equation: [(Total number of late adverse events in each category/total number of late patient years) x 100]. Late adverse events are events that occur ≥ 31 days post-implant through each subject's last follow-up visit or contact. Late patient years are calculated by totaling the amount of time the valve is implanted in the patient while participating in the trial and the count begins at ≥ 31 days post-implant through all subject's last follow-up visit or contact.
Time Frame: Events occurring ≥ 31 days and up through 8 years post-implant
Population: This outcome is reported for subjects who received an Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve.
Measure: Number; unit: Linearized rate percentage
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 329
Linearized rate percentage
  Thromboembolism | 2.0
  All bleeding events | 5.8
  All paravalvular leak | 0.3
  Endocarditis | 0.3

2. Primary Outcome: Primary Effectiveness Endpoints
Description: The primary effectiveness endpoint will be the percentage of subjects in NYHA functional classification I or II at 8 years post-implant.
Time Frame: 8 years post-implant
Population: This outcome is reported for subjects who received an Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve. Note that the number of participants analyzed is different from that in the participant flow as there was some missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 106
Participants | 93

3. Secondary Outcome: Percent of Early Adverse Events
Description: Total number of early adverse events, in each category, occurring within 30 days of procedure divided by the number of enrolled subjects times 100.
Time Frame: Events occurring within 30 days of procedure
Population: This outcome is reported for subjects who received an Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve.
Measure: Number; unit: percentage
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 329
percentage
  Thromboembolism | 2.1
  Valve Thrombosis | 0.0
  All Bleeding Events | 12.2
  Major bleeding | 9.4
  Endocarditis | 0.0
  Hemolysis | 0.0
  Structural Valve Deterioration | 0.0
  Non-Structural Valve Dysfunction | 1.5
  Reoperation | 0.9
  Explant | 0.9
  Death | 2.7

4. Secondary Outcome: Subject's Average Score on the EQ-5D - Quality of Life Questionnaire Over Time
Description: The EQ-5D is a standardized questionnaire that asks subjects to rate themselves (no problems, some problems, extreme problems) on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale ranges from a minimum of 0 and a maximum of 100. A lower number indicates the participants experiences more problems and a higher number indicates the participants experiences fewer problems.
Time Frame: 6 months post-implant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 214
units on a scale
  Baseline | 63.1 (20.7)
  6 months | 75.4 (17.8)

5. Secondary Outcome: Number of Late Adverse Events Divided by Late Patient Years (Expressed as a Percentage) for the Magna Mitral Valve Implanted Cohort
Description: as for outcome 1
Time Frame: Events occurring ≥ 31 days and up through 8 years post-implant
Population: This outcome is reported for subjects who received an Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve.
Measure: Number; unit: Linearized rate percentage
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 329
Linearized rate percentage
  Thromboembolism | 2.0
  Valve Thrombosis | 0.1
  All Bleeding Events | 5.8
  Major bleeding | 3.2
  Endocarditis | 0.3
  Hemolysis | 0.0
  Structural Valve Deterioration | 1.8
  Non-Structural Valve Dysfunction | 0.4
  Reoperation | 0.2
  Explant | 1.1
  Death | 5.3

6. Secondary Outcome: Subject's Average Mean Gradient Measurement
Description: Mean gradient is the average flow of blood through the mitral valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher value is considered worse, and a lower value is considered better but the value is dependent on the size and type of valve.
Time Frame: Baseline and 8 years post-implant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 175
mmHg
  Baseline | 8.03 (5.42)
  8 years: number analyzed (Participants) | 71
  8 years | 5.70 (2.85)

7. Secondary Outcome: Subject's Average Peak Gradient Measurement
Description: Peak gradient is the maximum value measured of flow of blood through the mitral valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher valve is considered worse, and a lower value is considered better, but the value is dependent on the size and type of valve.
Time Frame: Baseline and 8 years post-implant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 176
mmHg
  Baseline | 18.56 (9.63)
  8 years: number analyzed (Participants) | 73
  8 years | 14.57 (6.62)

8. Secondary Outcome: Subject's Average Effective Orifice Area (EOA) Measurement
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the mitral valve. Effective orifice area is evaluated by echocardiography over time. In general, a higher value is considered better, and a lower value is considered worse, but the value is dependent on the size and type of valve.
Time Frame: Baseline and 8 years post-implant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 110
cm^2
  Baseline | 1.39 (0.93)
  8 years: number analyzed (Participants) | 60
  8 years | 1.90 (0.67)

9. Secondary Outcome: Subject's Average Effective Orifice Area Index (EOAI) Measurement
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the mitral valve divided by the person's body surface area. Effective orifice area index is evaluated by echocardiography over time. In general, a higher value is considered better, and a lower value is considered worse, but the value is dependent on the size of the patient and the size and type of valve.
Time Frame: Baseline and 8 years post-implant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 110
cm^2/m^2
  Baseline | 0.73 (0.48)
  8 years: number analyzed (Participants) | 60
  8 years | 1.03 (0.38)

10. Secondary Outcome: Subject's Average Cardiac Output Measurement
Description: Cardiac output is the amount of blood the heart pumps through the circulatory system in a minute. Cardiac output is evaluated by echocardiography over time. Normal cardiac output in healthy volunteers over 60 years of age was reported between 3.1 and 6.4 liters per minute. In general, a higher value is considered better, and a lower value is considered worse.
Time Frame: Baseline and 8 years post-implant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 138
L/min
  Baseline | 4.70 (1.67)
  8 years: number analyzed (Participants) | 60
  8 years | 6.02 (1.52)

11. Secondary Outcome: Subject's Average Cardiac Index Measurement
Description: Cardiac index (CI) evaluated by echocardiography. Cardiac index is an assessment of the cardiac output value based on the patient's size. To obtain the cardiac index, divide the cardiac output by the person's body surface area (BSA). Cardiac Index is a useful marker of how well the heart is functioning as a pump by directly correlating the volume of blood pumped by the heart with an individual's body surface area. Normal cardiac output index in healthy volunteers over 60 years of age was reported between 1.1 and 3.2 L/min/m^2. In general, a higher value is considered better, and a lower value is considered worse, but the value is dependent on the size of the patient.
Time Frame: Baseline and 8 years post-implant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 98
L/min/m^2
  Baseline | 2.50 (0.86)
  8 years: number analyzed (Participants) | 55
  8 years | 3.32 (0.91)

12. Secondary Outcome: Subject's Average Left Ventricular Mass Regression
Description: Patients can experience an enlargement of the left ventricle (chamber) of their heart because it works harder with a defective heart valve. Left ventricular mass regression evaluates if the patient experiences a decrease in the size of the left ventricle (chamber) after the repair or replacement of their heart valve.
Time Frame: Baseline and 8 years post-implant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Device - CEP Mitral Valve
Number analyzed (Participants) | 193
grams
  Baseline | 213.21 (90.50)
  8 years: number analyzed (Participants) | 73
  8 years | 163.71 (54.50)

13. Secondary Outcome: Subject's Average Red Blood Cell Count
Description: The red blood cell (RBC) count is a test that measures the number of oxygen-carrying blood cells in your blood. The red blood cell count normal range for women is 4.2 to 5.4 10^6 cells/microliters and for men is 4.7 to 6.1 10^6 cells/microliters. A high red blood cell count may indicate that you have a condition that's preventing you from getting enough oxygen. A low RBC may be caused by an infection, or a medical condition related to anemia. In general, results either lower or higher than the normal range may indicate something is wrong.
Time Frame: 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 6-year, 7-year, and 8-year follow-up visits
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^6 cells/uL
Groups:
- Device - CEP Mitral Valve - 25mm; Device - CEP Mitral Valve - 27mm; Device - CEP Mitral Valve - 29mm; Device - CEP Mitral Valve - 31mm; Device - CEP Mitral Valve - 33mm: Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve
Arm/Group | Device - CEP Mitral Valve - 25mm | Device - CEP Mitral Valve - 27mm | Device - CEP Mitral Valve - 29mm | Device - CEP Mitral Valve - 31mm | Device - CEP Mitral Valve - 33mm
Number analyzed (Participants) | 76 | 117 | 81 | 39 | 16
10^6 cells/uL
  6 months: number analyzed (Participants) | 60 | 90 | 66 | 29 | 10
  6 months | 4.4 (0.6) | 4.4 (0.6) | 4.3 (0.6) | 4.3 (0.6) | 4.6 (0.5)
  1 year: number analyzed (Participants) | 52 | 90 | 60 | 28 | 10
  1 year | 4.4 (0.5) | 4.3 (0.5) | 4.4 (0.5) | 4.2 (0.6) | 4.6 (0.4)
  2 years: number analyzed (Participants) | 48 | 82 | 52 | 23 | 9
  2 years | 4.3 (0.5) | 4.4 (0.5) | 4.4 (0.6) | 4.3 (0.6) | 4.6 (0.3)
  3 years: number analyzed (Participants) | 40 | 74 | 50 | 22 | 8
  3 years | 4.3 (0.5) | 4.4 (0.5) | 4.4 (0.7) | 4.3 (0.7) | 4.6 (0.3)
  4 years: number analyzed (Participants) | 37 | 63 | 47 | 21 | 7
  4 years | 4.3 (0.5) | 4.4 (0.4) | 4.3 (0.5) | 4.4 (0.6) | 4.6 (0.3)
  5 years: number analyzed (Participants) | 27 | 55 | 38 | 15 | 6
  5 years | 4.4 (0.5) | 4.4 (0.5) | 4.3 (0.6) | 4.2 (0.8) | 4.5 (0.4)
  6 years: number analyzed (Participants) | 25 | 47 | 29 | 16 | 6
  6 years | 4.3 (0.6) | 4.4 (0.5) | 4.3 (0.6) | 4.3 (0.8) | 4.6 (0.4)
  7 years: number analyzed (Participants) | 18 | 31 | 22 | 15 | 6
  7 years | 4.5 (0.5) | 4.3 (0.6) | 4.2 (0.7) | 4.1 (0.8) | 4.6 (0.3)
  8 years: number analyzed (Participants) | 16 | 30 | 22 | 10 | 5
  8 years | 4.3 (0.6) | 4.4 (0.6) | 4.3 (0.6) | 4.1 (1.0) | 4.4 (0.4)

14. Secondary Outcome: Subject's Average White Blood Cell Count
Description: Laboratory analysis of White Blood Cell (WBC) count on blood drawn from subject; WBC fight infection. The normal reference range for WBC count is 4.5 to 10.0 10^3 cells/microliters. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 6-year, 7-year, and 8-year follow-up visits
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Device - CEP Mitral Valve - 25mm | Device - CEP Mitral Valve - 27mm | Device - CEP Mitral Valve - 29mm | Device - CEP Mitral Valve - 31mm | Device - CEP Mitral Valve - 33mm
Number analyzed (Participants) | 76 | 117 | 81 | 39 | 16
10^3 cells/uL
  6 months: number analyzed (Participants) | 60 | 90 | 66 | 29 | 10
  6 months | 6.9 (1.6) | 6.9 (1.7) | 7.2 (2.1) | 7.1 (2.2) | 6.7 (1.2)
  1 year: number analyzed (Participants) | 52 | 90 | 60 | 29 | 10
  1 year | 7.1 (2.0) | 6.9 (2.0) | 7.1 (1.8) | 7.5 (2.0) | 7.2 (1.3)
  2 years: number analyzed (Participants) | 48 | 82 | 52 | 23 | 9
  2 years | 6.9 (2.4) | 6.8 (1.9) | 7.2 (2.0) | 6.5 (1.8) | 5.8 (1.2)
  3 years: number analyzed (Participants) | 40 | 74 | 50 | 22 | 8
  3 years | 6.5 (2.4) | 6.8 (1.8) | 7.0 (2.2) | 7.1 (2.2) | 6.1 (1.3)
  4 years: number analyzed (Participants) | 37 | 62 | 47 | 21 | 7
  4 years | 6.9 (2.7) | 6.9 (1.9) | 7.6 (2.6) | 6.5 (1.6) | 6.0 (1.3)
  5 years: number analyzed (Participants) | 27 | 55 | 38 | 15 | 6
  5 years | 6.2 (1.7) | 6.8 (1.7) | 7.3 (2.2) | 6.8 (1.7) | 6.9 (3.8)
  6 years: number analyzed (Participants) | 25 | 47 | 29 | 16 | 6
  6 years | 6.4 (2.0) | 7.0 (1.6) | 6.9 (2.1) | 7.4 (1.8) | 5.9 (1.0)
  7 years: number analyzed (Participants) | 18 | 31 | 22 | 15 | 6
  7 years | 6.8 (2.3) | 7.2 (2.2) | 7.0 (2.2) | 6.7 (2.1) | 6.1 (1.7)
  8 years: number analyzed (Participants) | 16 | 30 | 22 | 10 | 5
  8 years | 6.0 (1.7) | 7.0 (2.1) | 7.9 (2.1) | 5.8 (1.5) | 6.6 (1.1)

15. Secondary Outcome: Subject's Average Hemoglobin Count
Description: This is the laboratory analysis of Hemoglobin count on blood drawn from subjects. Hemoglobin is an oxygen-carrying protein in red blood cells. In males, a healthy hemoglobin level is between 13.2 and 16.6 g/dL. In females, a hemoglobin count of between 11.6 and 15 g/dL is considered normal and healthy. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 6-year, 7-year, and 8-year follow-up visits
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Device - CEP Mitral Valve - 25mm | Device - CEP Mitral Valve - 27mm | Device - CEP Mitral Valve - 29mm | Device - CEP Mitral Valve - 31mm | Device - CEP Mitral Valve - 33mm
Number analyzed (Participants) | 76 | 117 | 81 | 39 | 16
g/dL
  6 months: number analyzed (Participants) | 60 | 90 | 66 | 29 | 10
  6 months | 12.4 (1.6) | 12.5 (1.5) | 12.8 (1.3) | 12.8 (1.6) | 13.7 (2.2)
  1 year: number analyzed (Participants) | 52 | 90 | 60 | 29 | 10
  1 year | 12.9 (1.5) | 12.8 (1.7) | 13.3 (1.4) | 12.9 (1.7) | 13.9 (1.4)
  2 years: number analyzed (Participants) | 48 | 82 | 52 | 23 | 9
  2 years | 12.5 (2.3) | 13.2 (1.4) | 13.3 (1.7) | 13.2 (1.9) | 14.0 (1.1)
  3 years: number analyzed (Participants) | 40 | 74 | 50 | 22 | 8
  3 years | 12.9 (1.5) | 13.0 (1.5) | 13.1 (1.4) | 13.1 (2.0) | 14.0 (1.8)
  4 years: number analyzed (Participants) | 37 | 62 | 47 | 21 | 7
  4 years | 12.6 (1.5) | 13.0 (1.5) | 12.9 (1.6) | 13.6 (1.7) | 14.2 (0.7)
  5 years: number analyzed (Participants) | 27 | 55 | 38 | 15 | 6
  5 years | 13.1 (1.4) | 13.0 (1.7) | 13.0 (1.6) | 13.0 (2.3) | 13.8 (1.4)
  6 years: number analyzed (Participants) | 25 | 47 | 29 | 16 | 6
  6 years | 12.5 (1.7) | 12.7 (1.7) | 12.7 (1.3) | 13.4 (2.0) | 14.4 (1.1)
  7 years: number analyzed (Participants) | 18 | 31 | 22 | 15 | 6
  7 years | 12.8 (1.6) | 12.7 (1.7) | 12.3 (1.8) | 12.7 (2.3) | 14.0 (1.5)
  8 years: number analyzed (Participants) | 16 | 30 | 22 | 10 | 5
  8 years | 12.5 (1.7) | 12.8 (2.0) | 13.1 (1.4) | 12.8 (2.7) | 13.6 (1.8)

16. Secondary Outcome: Subject's Average Hematocrit Count
Description: This is laboratory analysis of Hematocrit percentage on blood drawn from subjects. A hematocrit test measures the proportion of red blood cells in your blood. Red blood cells carry oxygen throughout your body. Having too few or too many red blood cells can be a sign of certain diseases. Normal hematocrit ranges for adult females are 36% to 44% and for adult males are 41% to 50%. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 6-year, 7-year, and 8-year follow-up visits
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Device - CEP Mitral Valve - 25mm | Device - CEP Mitral Valve - 27mm | Device - CEP Mitral Valve - 29mm | Device - CEP Mitral Valve - 31mm | Device - CEP Mitral Valve - 33mm
Number analyzed (Participants) | 76 | 117 | 81 | 39 | 16
Percentage of red blood cells
  6 months: number analyzed (Participants) | 60 | 90 | 66 | 29 | 10
  6 months | 38.0 (4.3) | 37.9 (4.3) | 38.7 (3.8) | 38.6 (4.8) | 40.7 (5.9)
  1 year: number analyzed (Participants) | 52 | 90 | 60 | 29 | 10
  1 year | 39.4 (4.0) | 38.6 (4.3) | 39.7 (4.1) | 38.6 (4.8) | 41.6 (3.6)
  2 years: number analyzed (Participants) | 48 | 82 | 52 | 23 | 9
  2 years | 39.0 (4.5) | 39.6 (3.7) | 40.0 (4.7) | 39.9 (5.1) | 41.6 (3.1)
  3 years: number analyzed (Participants) | 40 | 74 | 50 | 22 | 8
  3 years | 39.4 (4.4) | 39.1 (4.3) | 39.5 (3.8) | 39.4 (5.2) | 41.7 (5.0)
  4 years: number analyzed (Participants) | 37 | 62 | 47 | 21 | 7
  4 years | 39.0 (4.7) | 39.4 (3.9) | 39.2 (4.3) | 40.9 (4.3) | 42.4 (1.2)
  5 years: number analyzed (Participants) | 27 | 55 | 38 | 15 | 6
  5 years | 40.0 (4.5) | 39.7 (4.6) | 39.8 (4.7) | 39.4 (6.5) | 41.0 (3.7)
  6 years: number analyzed (Participants) | 25 | 47 | 29 | 16 | 6
  6 years | 38.7 (4.8) | 39.3 (4.6) | 38.8 (4.0) | 40.3 (5.9) | 42.3 (3.1)
  7 years: number analyzed (Participants) | 18 | 31 | 22 | 15 | 6
  7 years | 39.8 (4.8) | 37.3 (8.2) | 38.1 (5.1) | 38.1 (6.1) | 42.4 (4.4)
  8 years: number analyzed (Participants) | 16 | 30 | 22 | 10 | 5
  8 years | 38.6 (5.5) | 39.6 (5.1) | 39.8 (4.2) | 38.5 (7.4) | 40.9 (5.3)

17. Secondary Outcome: Subject's Average Reticulocytes Percentage Over Time
Description: Laboratory Analysis of reticulocytes on blood drawn from subjects. Reticulocytes are newly produced immature red blood cells; a reticulocyte blood test measures the amount of these cells in the blood. The reference range for reticulocytes is 0.5 - 2.6 % of red blood cells. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 6-year, 7-year, and 8-year follow-up visits
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | Device - CEP Mitral Valve - 25mm | Device - CEP Mitral Valve - 27mm | Device - CEP Mitral Valve - 29mm | Device - CEP Mitral Valve - 31mm | Device - CEP Mitral Valve - 33mm
Number analyzed (Participants) | 76 | 117 | 81 | 39 | 16
Percentage of reticulocytes
  6 months: number analyzed (Participants) | 60 | 87 | 63 | 28 | 9
  6 months | 1.2 (0.6) | 1.4 (0.7) | 1.4 (0.6) | 1.2 (0.6) | 1.1 (0.4)
  1 year: number analyzed (Participants) | 48 | 88 | 59 | 26 | 9
  1 year | 1.4 (0.6) | 1.4 (0.6) | 1.3 (0.5) | 1.3 (0.5) | 1.2 (0.6)
  2 years: number analyzed (Participants) | 46 | 80 | 49 | 23 | 8
  2 years | 1.5 (0.6) | 1.4 (0.5) | 1.4 (0.6) | 1.2 (0.4) | 2.9 (4.9)
  3 years: number analyzed (Participants) | 38 | 70 | 46 | 21 | 7
  3 years | 1.5 (0.5) | 1.5 (0.7) | 1.4 (0.5) | 1.3 (0.5) | 1.2 (0.6)
  4 years: number analyzed (Participants) | 34 | 63 | 43 | 21 | 7
  4 years | 1.4 (0.5) | 2.8 (10.3) | 1.6 (0.5) | 1.2 (0.4) | 1.1 (0.4)
  5 years: number analyzed (Participants) | 26 | 56 | 37 | 14 | 6
  5 years | 1.4 (0.5) | 2.6 (6.6) | 1.5 (0.6) | 1.4 (0.4) | 1.3 (0.5)
  6 years: number analyzed (Participants) | 25 | 45 | 28 | 14 | 6
  6 years | 1.5 (0.5) | 1.5 (0.6) | 1.4 (0.6) | 1.4 (0.4) | 1.1 (0.3)
  7 years: number analyzed (Participants) | 16 | 31 | 21 | 12 | 6
  7 years | 1.6 (0.4) | 2.0 (2.8) | 1.7 (1.0) | 1.3 (0.5) | 1.2 (0.2)
  8 years: number analyzed (Participants) | 16 | 29 | 19 | 8 | 4
  8 years | 1.6 (0.5) | 1.5 (0.6) | 2.2 (2.8) | 1.6 (0.8) | 1.5 (0.3)

18. Secondary Outcome: Subject's Average Platelet Count Over Time
Description: This is laboratory analysis of Platelet count on blood drawn from subjects. The purpose of platelets is to create hemostasis, which is the prevention of hemorrhaging (bleeding) and the process of keeping blood inside the vessel walls. A normal platelet range is 150 to 450 10^3 cells/microliter. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 6-year, 7-year, and 8-year follow-up visits
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | Device - CEP Mitral Valve - 25mm | Device - CEP Mitral Valve - 27mm | Device - CEP Mitral Valve - 29mm | Device - CEP Mitral Valve - 31mm | Device - CEP Mitral Valve - 33mm
Number analyzed (Participants) | 76 | 117 | 81 | 39 | 16
10^3 cells/microliter
  6 months: number analyzed (Participants) | 59 | 90 | 66 | 29 | 10
  6 months | 242.2 (85.7) | 218.5 (83.7) | 211.6 (68.9) | 202.0 (49.2) | 202.0 (58.4)
  1 year: number analyzed (Participants) | 51 | 90 | 60 | 29 | 10
  1 year | 224.3 (64.9) | 214.7 (76.9) | 201.6 (69.1) | 196.0 (42.1) | 201.5 (54.2)
  2 years: number analyzed (Participants) | 47 | 82 | 52 | 23 | 9
  2 years | 217.1 (66.8) | 208.9 (70.2) | 208.4 (80.5) | 190.6 (35.9) | 175.9 (31.0)
  3 years: number analyzed (Participants) | 39 | 74 | 50 | 22 | 8
  3 years | 208.0 (87.2) | 210.8 (80.2) | 200.3 (86.6) | 197.4 (45.8) | 191.0 (48.9)
  4 years: number analyzed (Participants) | 36 | 62 | 47 | 21 | 7
  4 years | 207.2 (79.7) | 212.0 (78.6) | 213.8 (108.2) | 188.1 (45.6) | 190.9 (40.3)
  5 years: number analyzed (Participants) | 26 | 55 | 38 | 15 | 6
  5 years | 203.5 (64.5) | 208.1 (74.6) | 207.4 (123.8) | 177.7 (37.6) | 212.2 (65.7)
  6 years: number analyzed (Participants) | 25 | 47 | 29 | 16 | 6
  6 years | 197.0 (61.3) | 214.3 (90.9) | 224.0 (197.2) | 190.4 (35.0) | 185.3 (27.3)
  7 years: number analyzed (Participants) | 17 | 31 | 22 | 15 | 6
  7 years | 203.4 (60.2) | 219.6 (77.3) | 237.2 (197.9) | 202.4 (46.7) | 181.5 (37.1)
  8 years: number analyzed (Participants) | 15 | 29 | 22 | 10 | 5
  8 years | 175.1 (48.4) | 225.1 (92.3) | 198.8 (53.6) | 189.3 (40.5) | 177.8 (27.9)

19. Secondary Outcome: Subject's Average Serum Lactate Dehydrogenase (LDH) Over Time
Description: The serum lactate dehydrogenase (LDH) test looks for signs of damage to the body's tissues. Normal levels of LDH in the blood can vary depending on the lab but usually range between 140 units per liter (U/L) to 280 U/L for adults and tend to be higher for children and teens. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 6-year, 7-year, and 8-year follow-up visits
Population: This outcome is reported for subjects who received an Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve. The protocol allowed subjects to have the option of having (haptoglobin and SLDH tests) or alternatively a plasma free hemoglobin test at each timeframe. Note that the number of participants analyzed is different from that in the participant flow as there was some missing data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Device - CEP Mitral Valve - 25mm | Device - CEP Mitral Valve - 27mm | Device - CEP Mitral Valve - 29mm | Device - CEP Mitral Valve - 31mm | Device - CEP Mitral Valve - 33mm
Number analyzed (Participants) | 76 | 117 | 81 | 39 | 16
U/L
  6 months: number analyzed (Participants) | 33 | 46 | 39 | 13 | 4
  6 months | 241.4 (48.4) | 247.3 (100.1) | 322.5 (189.8) | 274.2 (141.0) | 300.5 (182.0)
  1 year: number analyzed (Participants) | 22 | 46 | 33 | 13 | 3
  1 year | 232.7 (44.0) | 250.2 (100.4) | 294.5 (145.0) | 229.5 (103.1) | 472.3 (223.8)
  2 years: number analyzed (Participants) | 18 | 33 | 25 | 8 | 3
  2 years | 228.7 (54.0) | 231.9 (82.0) | 263.8 (103.1) | 209.1 (51.6) | 405.3 (219.8)
  3 years: number analyzed (Participants) | 10 | 24 | 20 | 6 | 2
  3 years | 243.1 (41.4) | 227.0 (66.0) | 274.7 (102.0) | 240.2 (56.4) | 332.5 (149.2)
  4 years: number analyzed (Participants) | 9 | 15 | 13 | 6 | 2
  4 years | 243.0 (53.1) | 220.1 (45.0) | 247.8 (33.7) | 251.0 (43.7) | 286.0 (127.3)
  5 years: number analyzed (Participants) | 4 | 10 | 11 | 2 | 2
  5 years | 227.3 (23.7) | 227.3 (42.5) | 221.4 (31.3) | 238.5 (19.1) | 287.0 (118.8)
  6 years: number analyzed (Participants) | 3 | 10 | 10 | 4 | 1
  6 years | 256.7 (71.3) | 248.5 (94.4) | 245.3 (33.8) | 269.3 (43.0) | 393
  7 years: number analyzed (Participants) | 0 | 6 | 6 | 4 | 1
  7 years |  | 202.5 (109.7) | 255.8 (24.2) | 254.0 (22.0) | 200.0
  8 years: number analyzed (Participants) | 1 | 4 | 5 | 3 | 1
  8 years | 253.0 | 254.5 (56.1) | 257.4 (28.4) | 369.7 (189.7) | 423.0

20. Secondary Outcome: Subject's Average Plasma Free Hemoglobin Over Time
Description: Laboratory analysis of Plasma Free Hemoglobin (Pf Hgb) of blood drawn from subject. This blood test measures the level of free hemoglobin in the plasma (liquid portion of the blood). The reference range for plasma free hemoglobin is 0.0 to 15.2 mg/dL. In general, values higher than this can indicate something is wrong.
Time Frame: 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 6-year, 7-year, and 8-year follow-up visits
Population: This outcome is reported for subjects who received an Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve. The protocol allowed subjects to have the option of having a plasma free hemoglobin test or alternatively a (haptoglobin and SLDH tests) at each timeframe. Note that the number of participants analyzed is different from that in the participant flow as there was some missing data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Device - CEP Mitral Valve - 25mm | Device - CEP Mitral Valve - 27mm | Device - CEP Mitral Valve - 29mm | Device - CEP Mitral Valve - 31mm | Device - CEP Mitral Valve - 33mm
Number analyzed (Participants) | 76 | 117 | 81 | 39 | 16
mg/dL
  6 months: number analyzed (Participants) | 25 | 39 | 24 | 11 | 5
  6 months | 10.7 (8.6) | 8.3 (7.2) | 14.4 (23.4) | 17.8 (35.3) | 20.1 (19.0)
  1 year: number analyzed (Participants) | 25 | 36 | 23 | 14 | 5
  1 year | 16.3 (17.5) | 11.7 (11.6) | 11.5 (13.5) | 18.3 (25.7) | 12.6 (8.0)
  2 years: number analyzed (Participants) | 27 | 43 | 23 | 13 | 3
  2 years | 15.2 (19.3) | 14.0 (18.4) | 7.9 (6.5) | 17.0 (14.0) | 12.3 (7.6)
  3 years: number analyzed (Participants) | 24 | 42 | 25 | 10 | 5
  3 years | 15.8 (20.1) | 11.6 (14.2) | 9.0 (8.7) | 7.4 (5.3) | 15.4 (8.9)
  4 years: number analyzed (Participants) | 21 | 42 | 29 | 11 | 4
  4 years | 26.3 (35.2) | 8.4 (7.5) | 13.6 (29.9) | 16.2 (21.8) | 10.0 (3.2)
  5 years: number analyzed (Participants) | 20 | 36 | 23 | 10 | 3
  5 years | 13.8 (17.6) | 7.5 (5.8) | 9.7 (9.5) | 9.6 (10.9) | 17.0 (7.8)
  6 years: number analyzed (Participants) | 18 | 28 | 15 | 8 | 5
  6 years | 14.0 (15.0) | 6.6 (4.1) | 12.2 (13.7) | 12.1 (11.9) | 29.8 (40.2)
  7 years: number analyzed (Participants) | 13 | 20 | 12 | 7 | 4
  7 years | 20.6 (32.1) | 12.3 (24.5) | 20.7 (31.5) | 8.5 (5.6) | 9.0 (4.8)
  8 years: number analyzed (Participants) | 12 | 21 | 11 | 5 | 4
  8 years | 14.2 (12.2) | 11.5 (9.7) | 12.5 (11.2) | 13.7 (11.8) | 8.0 (2.9)

21. Secondary Outcome: Subject's Average Haptoglobin Over Time
Description: Haptoglobin is a protein produced by your liver. It binds with hemoglobin, which is a protein found in red blood cells. When red blood cells are destroyed, they release hemoglobin. The released hemoglobin is called "free hemoglobin." Haptoglobin attaches to the free hemoglobin to create a haptoglobin-hemoglobin complex. This complex travels to the liver, where it's removed from the body. A normal haptoglobin level falls between 45 and 200 milligrams of haptoglobin per deciliter of blood. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: 6-month, 1-year, 2-year, 3-year, 4-year, 5-year, 6-year, 7-year, and 8-year follow-up visits
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Device - CEP Mitral Valve - 25mm | Device - CEP Mitral Valve - 27mm | Device - CEP Mitral Valve - 29mm | Device - CEP Mitral Valve - 31mm | Device - CEP Mitral Valve - 33mm
Number analyzed (Participants) | 76 | 117 | 81 | 39 | 16
mg/dL
  6 months: number analyzed (Participants) | 33 | 46 | 39 | 13 | 4
  6 months | 118.7 (59.0) | 143.9 (90.8) | 118.0 (63.6) | 119.2 (65.5) | 70.9 (68.4)
  1 year: number analyzed (Participants) | 22 | 45 | 31 | 13 | 3
  1 year | 110.0 (52.0) | 120.8 (68.9) | 107.9 (67.0) | 128.3 (60.5) | 123.7 (62.1)
  2 years: number analyzed (Participants) | 16 | 33 | 24 | 8 | 2
  2 years | 110.1 (38.9) | 127.1 (76.2) | 124.2 (57.6) | 101.8 (48.3) | 109.8 (89.4)
  3 years: number analyzed (Participants) | 12 | 23 | 18 | 7 | 2
  3 years | 103.6 (46.6) | 139.2 (80.3) | 96.2 (52.5) | 117.0 (36.1) | 109.0 (19.8)
  4 years: number analyzed (Participants) | 9 | 15 | 13 | 6 | 2
  4 years | 111.4 (54.9) | 139.9 (77.9) | 97.6 (49.6) | 96.9 (53.5) | 81.1 (113.0)
  5 years: number analyzed (Participants) | 4 | 9 | 10 | 2 | 2
  5 years | 79.0 (49.1) | 152.4 (81.5) | 111.6 (56.3) | 80.2 (91.6) | 120.1 (168.1)
  6 years: number analyzed (Participants) | 3 | 8 | 9 | 4 | 2
  6 years | 118.7 (95.5) | 109.8 (71.4) | 103.6 (58.6) | 126.8 (37.9) | 151.0 (70.7)
  7 years: number analyzed (Participants) | 0 | 5 | 6 | 4 | 1
  7 years |  | 85.2 (78.0) | 107.2 (72.6) | 51.7 (40.2) | 239.0
  8 years: number analyzed (Participants) | 1 | 3 | 5 | 2 | 1
  8 years | 115.0 | 129.0 (23.3) | 106.4 (40.0) | 96.0 (22.6) | 117.0

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through eight years of follow-up post implant.
Description: Adverse event table is reported for subjects who received the Carpentier-Edwards PERIMOUNT Magna Mitral surgical heart valve.
Arm/Group | Device - CEP Mitral Valve
All-Cause Mortality (participants affected / at risk) | 88/329
Serious Adverse Events (participants affected / at risk) | 281/329
Other Adverse Events (participants affected / at risk) | 206/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device - CEP Mitral Valve (N=329)
BLEEDING - MAJOR (Blood and lymphatic system disorders) | 60 (78)
BLEEDING - MINOR (Blood and lymphatic system disorders) | 23 (26)
ANGINA (Cardiac disorders) | 13 (19)
AORTIC REGURGITATION (NATIVE) (Cardiac disorders) | 2 (2)
ARRHYTHMIA (Cardiac disorders) | 99 (149)
CARDIAC CONDUCTION DISTURBANCE (Cardiac disorders) | 52 (52)
CARDIAC FAILURE (Cardiac disorders) | 73 (108)
CARDIOVASCULAR - OTHER (Cardiac disorders) | 32 (37)
CARDIOVASCULAR DISSECTION / TEAR / INJURY (Cardiac disorders) | 4 (4)
ENDOCARDITIS (Cardiac disorders) | 5 (5)
MYOCARDIAL INFARCTION (Cardiac disorders) | 6 (6)
NSVD - INAPPROPRIATE SIZING (Cardiac disorders) | 1 (1)
NSVD - PARAVALVULAR LEAK - MAJOR (Cardiac disorders) | 7 (7)
PLEURAL EFFUSION (Cardiac disorders) | 49 (57)
PNEUMOTHORAX / HEMOTHORAX (Cardiac disorders) | 3 (3)
PULMONARY EMBOLISM (Cardiac disorders) | 6 (6)
SVD - OTHER STRUCTURAL VALVE DETERIORATION (Cardiac disorders) | 10 (10)
SVD - STUDY VALVE CALCIFICATION (Cardiac disorders) | 6 (6)
SVD - STUDY VALVE WEAR (Cardiac disorders) | 1 (1)
THROMBOEMBOLISM - NON-CEREBRAL (Cardiac disorders) | 3 (4)
THROMBOEMBOLISM - STROKE (Cardiac disorders) | 18 (20)
THROMBOEMBOLISM - TIA (Cardiac disorders) | 6 (7)
TRICUSPID REGURGITATION (NATIVE) (Cardiac disorders) | 2 (2)
VALVE THROMBOSIS (Cardiac disorders) | 1 (1)
VASCULAR COMPLICATION (Cardiac disorders) | 11 (11)
VENTRICULAR RUPTURE (Cardiac disorders) | 2 (2)
ABNORMAL LAB VALUES (Blood and lymphatic system disorders) | 9 (11)
ANEMIA (Blood and lymphatic system disorders) | 31 (32)
BONE FRACTURE (Musculoskeletal and connective tissue disorders) | 29 (32)
CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 (33)
CARDIAC ARREST (Cardiac disorders) | 8 (9)
COAGULOPATHY (Blood and lymphatic system disorders) | 5 (5)
DRUG REACTION (General disorders) | 2 (2)
EDEMA (General disorders) | 3 (3)
FEVER - UNKNOWN ORIGIN (Infections and infestations) | 1 (1)
GASTRO-INTESTINAL COMPLICATION (Gastrointestinal disorders) | 53 (69)
HEMATOLOGICAL DISORDER (Blood and lymphatic system disorders) | 19 (21)
HEPATIC COMPLICATION (Hepatobiliary disorders) | 6 (6)
HYPERTENSION (General disorders) | 5 (6)
HYPOTENSION (General disorders) | 5 (5)
INFECTION / INFLAMMATION (Infections and infestations) | 59 (98)
METABOLIC COMPLICATION (Metabolism and nutrition disorders) | 11 (11)
MULTIPLE ORGAN FAILURE (General disorders) | 12 (12)
NEUROLOGICAL COMPLICATION (General disorders) | 18 (20)
OTHER (General disorders) | 79 (112)
PSYCHIATRIC COMPLICATION (Psychiatric disorders) | 10 (10)
RENAL COMPLICATION (Renal and urinary disorders) | 36 (42)
RESPIRATORY COMPLICATION (Respiratory, thoracic and mediastinal disorders) | 86 (133)
SEPTICEMIA (General disorders) | 10 (11)
STERNAL / THORACIC WOUND COMPLICATION (General disorders) | 11 (11)
SUDDEN DEATH (General disorders) | 5 (5)
SUICIDE (General disorders) | 1 (1)
SYNCOPE (General disorders) | 12 (13)
URINARY TRACT INFECTION (Renal and urinary disorders) | 12 (15)
VISION DISORDER (Eye disorders) | 11 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device - CEP Mitral Valve (N=329)
BLEEDING - MINOR (Blood and lymphatic system disorders) | 17 (22)
ARRHYTHMIA (Cardiac disorders) | 70 (108)
CARDIAC CONDUCTION DISTURBANCE (Cardiac disorders) | 34 (42)
CARDIOVASCULAR - OTHER (Cardiac disorders) | 26 (32)
PLEURAL EFFUSION (Cardiac disorders) | 44 (45)
ABNORMAL LAB VALUES (Blood and lymphatic system disorders) | 26 (41)
ANEMIA (Blood and lymphatic system disorders) | 36 (40)
GASTRO-INTESTINAL COMPLICATION (Gastrointestinal disorders) | 24 (30)
HEMATOLOGICAL DISORDER (Blood and lymphatic system disorders) | 27 (30)
HYPOTENSION (General disorders) | 18 (22)
INFECTION / INFLAMMATION (Infections and infestations) | 35 (54)
NEUROLOGICAL COMPLICATION (General disorders) | 19 (24)
OTHER (General disorders) | 78 (173)
RENAL COMPLICATION (Renal and urinary disorders) | 31 (34)
RESPIRATORY COMPLICATION (Respiratory, thoracic and mediastinal disorders) | 62 (96)
URINARY TRACT INFECTION (Renal and urinary disorders) | 30 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of overall study results which have not been released requires written approval of Sponsor, but presentation of site-specific results can occur subject to review by Sponsor. Manuscripts will be submitted to Sponsor for review 30 days prior to submission of manuscript for publication/presentation. Sponsor may ask for a 60-day delay of submission of manuscripts for publication to protect proprietary information and filing of related patent applications.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-11-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT00853632/Prot_SAP_ICF_000.pdf